CLINICAL TRIAL: NCT04268641
Title: Evaluation of Positioning Protocols with an Adapted Equipment on a Wheelchair in Hemiplegic Patients Following a Stroke
Brief Title: Evaluation of Positioning Protocols on a Wheelchair in Hemiplegic Patients
Acronym: POSIT-HEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: GHIV0417
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Hemiplegia And/or Hemiparesis Following Stroke
Keywords: Hemiplegia; Stroke; Wheelchair positioning; Propulsion; Pelvic posterior tilt; Obliquity
MeSH Terms: conditions — Hemiplegia; Stroke | interventions — DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Use of positioning equipment order 1 (Experimental): One standardized course is performed 3 times by each patient : one with a standard wheelchair and the 2 other with one or two positioning equipment (Seat back or/and positioning cushion) Each arm differs from the previous by the order of use of the equipment.
  Interventions: Other: Arm 1
- Use of positioning equipment order 2 (Experimental): One standardized course is performed 3 times by each patient : one with a standard wheelchair and the 2 other with one or two positioning equipment (Seat back or/and positioning cushion) Each arm differs from the previous by the order of use of the equipment.
  Interventions: Other: Arm 2
- Use of positioning equipment order 3 (Experimental): One standardized course is performed 3 times by each patient : one with a standard wheelchair and the 2 other with one or two positioning equipment (Seat back or/and positioning cushion) Each arm differs from the previous by the order of use of the equipment.
  Interventions: Other: Arm 3
- Use of positioning equipment order 4 (Experimental): One standardized course is performed 3 times by each patient : one with a standard wheelchair and the 2 other with one or two positioning equipment (Seat back or/and positioning cushion) Each arm differs from the previous by the order of use of the equipment.
  Interventions: Other: Arm 4
- Use of positioning equipment order 5 (Experimental): One standardized course is performed 3 times by each patient : one with a standard wheelchair and the 2 other with one or two positioning equipment (Seat back or/and positioning cushion) Each arm differs from the previous by the order of use of the equipment.
  Interventions: Other: Arm 5
- Use of positioning equipment order 6 (Experimental): One standardized course is performed 3 times by each patient : one with a standard wheelchair and the 2 other with one or two positioning equipment (Seat back or/and positioning cushion) Each arm differs from the previous by the order of use of the equipment.
  Interventions: Other: Arm 6

INTERVENTIONS:
Other: Arm 1 — Materials used for the course :
  1. : Standard Wheelchair
  2. : Standard Wheelchair + Seat back + Positioning cushion
  3. : Standard Wheelchair + Seat back + Positioning cushion + Belt
  Arms: Use of positioning equipment order 1
Other: Arm 2 — Materials used for the course :
  1. : Standard Wheelchair
  2. : Standard Wheelchair + Seat back + Positioning cushion + Belt
  3. : Standard Wheelchair + Seat back + Positioning cushion
  Arms: Use of positioning equipment order 2
Other: Arm 3 — Materials used for the course :
  1. : Standard Wheelchair + Seat back + Positioning cushion
  2. : Standard Wheelchair + Seat back + Positioning cushion + Belt
  3. : Standard Wheelchair
  Arms: Use of positioning equipment order 3
Other: Arm 4 — Materials used for the course :
  1. : Standard Wheelchair + Seat back + Positioning cushion
  2. : Standard Wheelchair
  3. : Standard Wheelchair + Seat back + Positioning cushion + Belt
  Arms: Use of positioning equipment order 4
Other: Arm 5 — Materials used for the course :
  1. : Standard Wheelchair + Seat back + Positioning cushion + Belt
  2. : Standard Wheelchair
  3. : Standard Wheelchair + Seat back + Positioning cushion
  Arms: Use of positioning equipment order 5
Other: Arm 6 — Materials used for the course :
  1. : Standard Wheelchair + Seat back + Positioning cushion + Belt
  2. : Standard Wheelchair + Seat back + Positioning cushion
  3. : Standard Wheelchair
  Arms: Use of positioning equipment order 6

SUMMARY:
The main purpose of this study is to assess the interest of using wheelchair positioning equipment on the decrease of postural disorders, compared to the standard use of a wheelchair

DETAILED DESCRIPTION:
The stroke is the main cause of hemiplegia in developed countries. Fifteen percent of people who say they have a stroke need, at home, a wheelchair to get from one room to another. The use of a wheelchair can cause postural disorders which can lead to pain, orthopedic deformity and pressure ulcers.

This study aims to assess the interest of using wheelchair positioning equipment (Seat back, Positioning cushion and Belt) on the decrease of postural disorders.

This decrease will be assessed after a standardized course, performed under three different conditions: with the positioning equipment (Positioning cushion and Seat back), with the positioning equipment and the belt and with the wheelchair alone.

Clinical tool used to assess the decrease is the Seated Postural Control Measure for Adults 2.0 (SPCMA 2.0).

This study, which will be the first prospective, interventional, multicenter, controlled and randomized study, could pave the way for guidelines of good practice, for wheelchair positioning of hemiplegic patients in France

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patient following a stroke
* Hospitalized in a follow-up and rehabilitative care service, after hospital stays in a MCO service (neurology, neurosurgery or reanimation)
* With a planned exit from hospital (homecoming, residential care facilities, nursing home, Long Term Care Unit …)
* Patient whose wheelchair choice should be already done
* Patient who propels the wheelchair with the valid hand and/or valid foot
* Written informed consent (IC) obtained
* Patients with affiliation to the social security system

Exclusion Criteria:

* Good walk recovery (FAC scale >3)
* Wheelchair with a double hand rim
* Patient who cannot use his2 wheelchair independently
* Cognitive disorders which prevent the ability to well understanding the instructions
* Other pathology which can interfere with this protocol (Spinal disorder, morbid overweight (BMI>40…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Degree of pelvic posterior tilt | Immediately after the end of the procedure, an average of 1 day
  The Primary Outcome Measure is the variation of the Degree of pelvic posterior tilt at the end of the three standardized course. These courses were performed with Standard Wheelchair, Standard Wheelchair + Seat back + Positioning cushion + Belt or with Standard Wheelchair + Seat back + Positioning cushion.
  The Degree of pelvic posterior tilt was measured using the SPCMA 2.0 score (0 = normal, 1 = mild, 2 = moderate and 3 = severe retroversion)

SECONDARY OUTCOMES:
Variation of Degree of pelvic posterior tilt | Baseline and immediately after the end of the procedure, an average of 1 day
  The variation of the Degree of pelvic posterior tilt was measured between the beginning and the end of the three standardized course using the SPCMA 2.0 score (0 = normal, 1 = mild, 2 = moderate and 3 = severe retroversion)
Variation of degree of lateral inclination of the torso | Baseline and immediately after the end of the procedure, an average of 1 day
  The variation of the degree of lateral inclination of the torso was measured between the beginning and the end of the three standardized course using the SPCMA 2.0 score (0 = normal, 1 = mild, 2 = moderate and 3 = severe retroversion)
Variation of the degree of Pelvis obliquity | Baseline and immediately after the end of the procedure, an average of 1 day
  The variation of the degree of Pelvis obliquity was measured at the end of the three standardized course using the SPCMA 2.0 score (0 = normal, 1 = mild, 2 =moderate and 3 = severe retroversion)
Degree of lateral inclination of the torso | Immediately after the end of the procedure, an average of 1 day
  The degree of lateral inclination of the torso was measured at the end of the three standardized course using the SPCMA 2.0 score (0 = normal, 1 = mild, 2 = moderate and 3 = severe retroversion)
Degree of Pelvis obliquity | Immediately after the end of the procedure, an average of 1 day
  The degree of Pelvis obliquity was measured at the end of the three standardized course using the SPCMA 2.0 score (0 = normal, 1 = mild, 2 = moderate and 3 = severe retroversion)
Measure of patient's satisfaction | Immediately after the end of the procedure, an average of 1 day
  The satisfaction of patient was measured with a satisfaction questionnaire scale based on ease of movement, wheelchair comfort and pain during the course. For each item, patient ticks : Very satisfied, Satisfied, Neither satisfied or unsatisfied, Unsatisfied or Very unsatisfied
Ability to achieve the whole course | Immediately after the end of the procedure, an average of 1 day
  Binary criteria (Yes / No)
Adverse event collect | Immediately after the end of the procedure, an average of 1 day
  Total number of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Pellegrini, Principal Investigator — Groupement Hospitalier Intercommunal du Vexin
Locations (7):
- France (7):
  - Groupement Hospitalier Intercommunal du Vexin, Aincourt
  - Hôpital Raymond Poincaré, Garche
  - Institut Régional de Réadaptation, Lay-Saint-Christophe
  - Centre de l'ESPOIR, Lille
  - Centre de Rééducation L'oiseau Blanc, Mantes-la-Jolie
  - Centre de Rééducation et de Réadaptation Fonctionnelles, Menucourt
  - Centre Hospitalier Universitaire de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No